CLINICAL TRIAL: NCT03064516
Title: Endocrowns vs.Ceramic Onlays With Filling and Fiber Pins Used in Endodontically Treated Teeth- Randomized Clinical Study
Brief Title: Endocrowns vs.Ceramic Onlays Used in Endodontically Treated Teeth- Randomized Clinical Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Susana Morimoto (Other)
Responsible Party: Sponsor-Investigator, Susana Morimoto, Clinical Professor, Universidade Ibirapuera
Organization: Universidade Ibirapuera (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UNIB2
Record Dates: First submitted 2017-02-22; First posted 2017-02-27 (Actual); Last update posted 2019-10-30 (Actual); Status verified 2019-10

CONDITIONS: Ceramic Restorations in Endodontically Treated Teeth
MeSH Terms: interventions — Inlays

STUDY DESIGN:
Intervention Model Description: Two arms: Endocrowns vs partial ceramic restoration with post
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Endocrown (Experimental): Restorations with ceramic endocrown in endodontically treated teeth
  Interventions: Procedure: Endocrown
- Onlay and fiber pin (Active Comparator): Restorations with onlay ceramic and glass fiber pin in endodontically treated teeth
  Interventions: Procedure: Onlay and fiber pin

INTERVENTIONS:
Procedure: Endocrown — In experimental group, the researches will be performed in the Endocrown group- only the ceramic restoration will fill the pulp chambre in teeth treated endodontically. Cusps will be preserved.
  Arms: Endocrown
Procedure: Onlay and fiber pin — In control group, the researches will be performed in the onlay ceramic restorations with glass fiber pin group in endodontically treated teeth- the teeth receive a fiberglass pin in the main root canal and composite resin filling. Cusps will be preserved.
  Arms: Onlay and fiber pin

SUMMARY:
Objective: To evaluate the immediate and mediate outcomes of endocrowns and onlay ceramic restorations with glass fiber pin in endodontically treated teeth. Material and methods: A randomized controlled clinical trial, a double-blind (patient and examiner) is conducted by one trained and calibrated operators who perform all restorative procedures. The restorations are evaluated longitudinally by a blind and calibrated examiner using the USPHS. A total of 20 patients will be randomly assigned to each group for a total of 40 patients. The randomization sequence will be generated (www.sealedenvelope.com) and to ensure the confidentiality of the allocation, this will be used opaque, sealed and numbered envelopes in series. These will be kept with an independent researcher for the moment of inclusion of the subjects. In the group of onlays, the teeth receive a fiberglass pin in the main root canal and composite resin filling. In the group of endocrown, only the restoration fill the pulp chamber. The parts are milled in IPS e-max CAD (Ivoclar Vivadent) and cemented with the Multilink cementation system (Ivoclar Vivadent). The immediate clinical (focused in restoration and patient) and mediate (radiographic and clinical) outcomes will be compared between the groups. Survival and success rates will be defined in 24 months. Survival will be established by Kaplan-Meier survival curve and log-rank can be conducted to identify as variables associated with as failures over time. Multivariate analysis with the Cox regression models will be condutcted for the determination of failure predictors. For all analyzes, the significance value will be adjusted to 5%.

DETAILED DESCRIPTION:
Study design - ethical and methodological aspects This study is an integral part of an umbrella project, in which the primary outcome is the longevity of prosthetic treatments, whereas patient-centered secondary outcomes are dealt with in the current study. The study protocol was approved by the Research Ethics Committee, following the Consolidated Standards of Reporting of Trials (CONSORT and CONSORT PRO) guidelines (Calvert et al., 2013; Moher et al., 2012), and registered at clinicaltrials.gov (NCT03064516).

This double-blind, parallel-arm randomized clinical trial, with a 1:1 allocation ratio, was conducted by a previously trained operator, who performed all the restorative procedures.

Survival rate of inlay/onlay ceramic restorations (96.6% after 24 months) was the primary outcome considered for sample size calculation (Peumans et al., 2010). Therefore, a clinically significant difference of 15% is expected for longevity between the groups. So, adopting a significance level of 0.05 and a 0.80 power, considering one tooth per patient, and using a two-tailed test for noninferiority trials, adding 20% for possible losses (dropout), the final number of teeth per group was 20, corresponding to a total of 40 teeth.

Participants - recruitment, eligibility, randomization, and allocation The patients were recruited by one of the researchers (SM) based on history-taking, clinical examination, and radiographic exams using a sample of patients from the Military Police Dental Center (São Paulo, Brazil) treated in 2017. The clinical steps were carried out in a private dental office.

Eligible patients were randomly assigned to one of the parallel arms of the study. The randomization sequence was generated (www.sealedenvelope.com) and allocation concealment was ensured by the use of sealed brown envelopes numbered serially and kept in possession of an independent researcher until they were opened by the operator at the beginning of treatment. The contents of the envelope indicated the experimental group to which the patient would be assigned: Endocrown group (test) or Partial coverage ceramic restoration + fiber post group (PCCR+post- control).

Restorative techniques for the experimental groups All participants received instructions on oral hygiene and diet. Radiographs were taken at baseline and after cementation. Photographs were taken at baseline, after removal of the carious tissue and of old restorations, after cavity preparation, and after cementation. Procedure time was recorded in sessions 1 and 2, beginning with preoperative mouth rinsing and ending with occlusal adjustment (session 1) and beginning with preoperative mouth rinsing and ending with final radiograph (session 2).

Session 1- Cavity preparation and casting Endocrown group- Well-defined cervical chamfered finish lines should be created to facilitate the impression and technical procedures, thus a 2-mm round-ended chamfer finish line was created along the margin using tapered inverted cone diamond burs, at high rotation and under cooling, against a 1:5 contra angle multiplier (S-MAX M95L- NSK). No filling was used, the space of the pulp chamber is included in the preparation.

PCCR+Post group- A fiber post (White post, FGM) whose size was compatible with the main canal was luted, reaching approximately half of the canal. The post was cleaned with alcohol, dried, and treated with Monobond (Ivoclar Vivadent); Multilink was applied to the tooth (Ivoclar Vivadent), mixing it with primer A+B at a 1:1 ratio, without previous acid etching, with a brief air jet. After that, the post was luted with Multilink resin cement (Ivoclar Vivadent), followed by photopolymerization for 20 seconds and filling with composite resin - shade A2 (Tetric N Ceram bulk fill- Ivoclar Vivadent), in 1-2 mm increments and photopolymerization for 20 seconds per layer. Occlusal and proximal boxes were prepared, not exceeding 2 mm in ceramic thickness. A 2-mm round-ended chamfer finish line was created along the margin of extracoronal areas using tapered inverted cone diamond burs, at high rotation and under cooling, against a 1:5 contra angle multiplier (1:5 S-Max M95L, NSK).

In both groups, the cusps were preserved, whenever possible, but in cases where veneering was needed, the occlusal surface was abraded to allow for a 1.5-to-2 mm space. If necessary, the proximal contact point was removed with metal files.

The double-cord technique (Ultrapack- Ultradent) and double molding technique were used (Virtual heavy and regular body - Ivoclar Vivadent). The color was chosen using the Vita classical shade guide (Vita Zahnfabrik). The provisional restorations were fabricated with acrylic resin and cemented with Temp Bond NE (Kerr Corporation).

Laboratory phase - ceramic restoration manufacture The specimens were fabricated with lithium disilicate glass ceramic (IPS e.max CAD- Ivoclar Vivadent) and milled (Cerec In Lab Mcxl), producing a monolithic restoration, which was tinted and glazed.

Session 2- Testing, fitting, and cementation of the ceramic restoration After testing and fitting of the specimen in the mouth, rubber dam isolation was used for adhesive cementation in both groups, as follows: the enamel and dentin were etched with 37% phosphoric acid gel (N-etch; Ivoclar Vivadent) for 15-20 seconds, followed by copious rinsing and brief air jets. The specimens were etched with 5% hydrofluoric acid (IPS Ceramic Etching Gel; Ivoclar Vivadent), silanized for 1 min (Monobond N; Ivoclar Vivadent) and luted with Tetric N-bond and Multilink N dual cement (Ivoclar Vivadent). Photoactivation was performed with a Radii-Cal device (SDI- 1200 mW/cm2) for 20 seconds on each surface. Occlusal adjustment was performed and the restorations were polished with rubber points (Optra Fine Ivoclar Vivadent) at low speed, under cooling.

Patient-centered outcomes

Endodontic treatments had been carried out by different dentists on dates that could not be clearly specified by the patients. Patient-reported outcome measures (PROMs) include self-administered questionnaires, with the purpose of evaluating psychometric data, in addition to history taking and demographic and clinical data. The questionnaires described next were handed out to participants by an external examiner, in the absence of the operator:

* Patient satisfaction questionnaire (Mattos-Silveira et al., 2015) - The patient was asked to give his/her real opinion about the treatment and to indicate how satisfied he/she was on a 0-3 scale: 0 - excellent; 1- good; 2- acceptable; 3- not satisfied.
* Visual analog scale- Used to assess patient discomfort/pain immediately after the end of sessions 1 and 2. This scale consists of a 10-cm (100-mm) horizontal line, with "no sensitivity" written on one end and "maximum sensitivity" on the other one. The patient was asked to draw a vertical line on the horizontal scale to indicate his/her level of discomfort/pain. After that, the distance (in mm) from the starting point (no sensitivity) to the vertical line drawn by the patient was measured with a ruler (0 to 100 mm). The recorded values were interpreted as follows: 0-4 mm no discomfort; 5-44 mm mild discomfort; 45-74 mm moderate discomfort; 75-100 maximum discomfort.

Statistical analysis The data were assessed by SPSS V16 for Windows (SPSS; Chicago, IL, USA). Poisson regression analysis was used to compare patient discomfort between the groups and to evaluate the influence of explanatory variables on the discomfort reported by patients (age and sex, tooth, type of restorative treatment, number of treated surfaces, presence of endodontic lesion, and procedure time). At first, an unadjusted Poisson regression analysis was performed for each explanatory variable, and values with p<0.20 were included in the adjusted regression model. Only those variables with p=0.05 were kept in the final model. Prevalence ratios (PR) were calculated using a 95% confidence interval (95%CI). As the level of satisfaction was 100% for score 0, it was not possible to conduct a statistical analysis. Two-way repeated-measures analysis of variance - experimental group and time - was used to estimate the difference in procedure time between the experimental groups. Kaplan Meyer will be performed to survival analysis.

In all analyses, the significance level was set at 5%.

ELIGIBILITY:
Inclusion Criteria:

1. Presence of molars or pre molars with endodontic treatment with at least 1 face (buccal or lingual) or 1 cusp with adequate thickness of 3 mm;
2. Presence of opposing teeth and normal occlusion;
3. Supragingival margin after preparation;
4. Volunteers with good oral hygiene (no active caries, gingivitis, periodontal disease or any other disease in the soft or hard tissues of the oral cavity);
5. The selected teeth should not present restorations, cracks, hypoplasias or caries lesions in the adjacent remaining faces;
6. Not being in orthodontic treatment;
7. Be at least 18 years old.

Exclusion Criteria:

1. Patients will be excluded with special needs, using orthodontics devices and / or systemic diseases which may affect the oral cavity;
2. Teeth that undergo radiographic or clinical examination with painful symptomatology, unsatisfactory endodontic treatment, mobility, presence of abscess or fistula next to the tooth, teeth with restorations, sealants or enamel formation defects or signs of periapical alteration will also be excluded;

4) Volunteers smokers and pregnant women; 5) Volunteers without agenda compatible with the research schedule.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-03-20 (Actual); Primary Completion 2017-12-20 (Actual); Study Completion 2017-12-20 (Actual)

PRIMARY OUTCOMES:
Survival of restorations | Up to 24 months
  To evaluate the survival of different restorative treatments.

SECONDARY OUTCOMES:
Scale to discomfort | Immediately to restoration procedure
  Evaluate the discomfort of different restorative treatments
Cost-efficacy analysis by total value of treatment in relation to efficacy | Up to 24 months
  To evaluate the costs of different restorative treatments by total value in dollar of treatment in relation to efficacy. The researchers would like to analyze that a treatment of low cost show the similar efficacy of a high cost treatment.
Questionnaire of Oral health quality of life (OHIP) | Up to 24 months
  To evaluate the impact of different restorative treatments in oral health quality of life of patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidade Ibirapuera, São Paulo, São Paulo, Brazil